CLINICAL TRIAL: NCT04007224
Title: Comparison of Umbilical Cord Blood vs Personalized Treatment for Improving Autistic Spectrum Disorder
Brief Title: Umbilical Cord Blood vs Personalized Treatments for Improving Autistic Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundatia Bio-Forum (Other)
Collaborators: Spitalul Angiomedica (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORDUS
Record Dates: First submitted 2019-01-28; First posted 2019-07-05 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Autistic Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): Intranasal Oxytocin
  Interventions: Drug: Intranasal oxytocin
- Autologous umbilical cord blood (Experimental): Intravenous administration of autologous umbilical cord blood
  Interventions: Biological: Autologous umbilical cord blood

INTERVENTIONS:
Drug: Intranasal oxytocin — daily administration of oxytocin, 10 UI intrnasal, 5 UI bid, and if needed curcumin orally 250 mg bid, and/or lecithin 500 mg bid, and/or pironoquinolinquinone, 20 mg qd
  Other Names: non-invasive treatment
  Arms: Oxytocin
Biological: Autologous umbilical cord blood — patients aged between 3 and 7 years will receive one-time intravenously the processed umbilical cord blood collected at the respective child's birth
  Other Names: invasive treatment
  Arms: Autologous umbilical cord blood

SUMMARY:
The clinical study evaluates in an open-label, crossover design the comparative efficacy and safety of intranasal oxytocin and autologous umbilical cord blood for improving the functioning of children with autistic spectrum disorder

DETAILED DESCRIPTION:
Children aged 3-7 years diagnosed with autistic spectrum disorder and who did not previously receive oxytocin or umbilical cord blood treatments, will be enrolled to receive both treatments in random order. Assessment of functioning impairment will be done with QCHAT/M-CHAT/CAST questionnaires initially, at 2 months, 6 months and 1 year after first treatments. Either oxytocin or cord blood will be administered initially and at visit 2, which will take place at 2 months. All children will receive both treatments. A total of 25-40 children are expected to enroll and complete the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autistic spectrum disorder

Exclusion Criteria:

* metabolic or genetic disorder (ex storage disease, Down, etc),

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Improvement in behaviour, interaction with family and peers | At 2 months after administration of either treatment
  change in scores on M-CHAT (Modified Checklist for Autism in Toddlers) questionnaire; total score, maximum 20, lower is better
Improvement in behavior and social interaction | At 2 months after administration of either treatment
  change in score on Q-CHAT (Quantitative Checklist for Autism in Toddlers) questionnaire; total score, maximum 100, lower is better
Improvement in overall functioning of the child | At 2 months after administration of either treatment
  change in score on CAST (The Childhood Autistic Spectrum Test) questionnaire; Total score, maximum 39, lower is better

CONTACTS AND LOCATIONS:
Overall Officials: Felician Stancioiu, M.D., Principal Investigator — Fundatia Bio-Forum
Locations (2):
- Romania (2):
  - Spitalul Angiomedica, Bucharest, București
  - Medicover Hospital, Bucharest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stancioiu F, Bogdan R, Bulumac B, Ivanescu B, Dumitrescu R. Decontamination of Two Umbilical Cord Blood Grafts Prior to Autologous Administration. Maedica (Bucur). 2022 Dec;17(4):885-892. doi: 10.26574/maedica.2022.17.4.885. PMID 36818273

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT04007224/Prot_SAP_ICF_002.pdf